CLINICAL TRIAL: NCT03151005
Title: Randomized Clinical Trial to Evaluate The Effect of Metformin-GLP-1 Receptor Agonist Versus Oral Contraceptive (OC) Therapy on Reproductive Disorders and Cardiovascular Risks in Overweight Polycystic Ovarian Syndrome (PCOS) Patients
Brief Title: The Effect of GLP-1 Agonists Versus OCs on Reproductive Disorders and Cardiovascular Risks in Overweight PCOS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xinqiao Hospital of Chongqing (Other)
Responsible Party: Principal Investigator, Long Min,MD, Deputy Chief Physician, Associated professor, Xinqiao Hospital of Chongqing
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Xinqiao Endocrinology
Record Dates: First submitted 2017-04-28; First posted 2017-05-12 (Actual); Results first posted 2023-12-04 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Polycystic Ovary Syndrome (PCOS); Overweight; Obesity
Keywords: Polycystic Ovary Syndrome (PCOS); Overweight; Obesity; GLP-1 Agonist; Oral contraceptives (OCs); Metformin; Reproductive Disorders; Cardiovascular risk factor; Lipid Metabolism
MeSH Terms: conditions — Polycystic Ovary Syndrome; Overweight; Obesity | interventions — Metformin; Cyproterone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Metformin-GLP-1 Receptor Agonist (Experimental): Metformin-GLP-1 Receptor Agonist Therapy: metformin 0.5 g/time by mouth, 3 times per day, with 5 ug exenatide subcutaneous injection twice per day, for 4 weeks, then change to 10ug exenatide subcutaneous injection twice per day for 8 weeks; or metformin 0.5 g/time by mouth, 3 times per day, with 0.6mg liraglutide subcutaneous injection once per day, for 1 weeks, then change to 1.2-1.8 mg liraglutide subcutaneous injection according to patient's blood glucose condition, twice per day for 8 weeks.
  Interventions: Drug: Metformin-GLP-1 Receptor Agonist
- Metformin-Oral Contraceptive(OC) (Active Comparator): Metformin-Oral Contraceptive(OC) Therapy: metformin 0.5 g/ time by mouth, 3 times per day, with Diane 35(OC) 1 piece per day by mouth, for 12 weeks.
  Interventions: Drug: Metformin-Oral Contraceptive(OC)

INTERVENTIONS:
Drug: Metformin-GLP-1 Receptor Agonist — metformin oral with exenatide/liraglutide subcutaneous injection.
  Other Names: Metformin-exenatide/liraglutide Therapy
  Arms: Metformin-GLP-1 Receptor Agonist
Drug: Metformin-Oral Contraceptive(OC) — metformin with Diane 35 oral intake.
  Other Names: Metformin, Diane 35
  Arms: Metformin-Oral Contraceptive(OC)

SUMMARY:
Polycystic ovary syndrome (PCOS) is a health problem that affects one in 10 women of childbearing age, which is usually characterized by hormonal imbalance and metabolism problems such as hyperandrogenism and obesity. Diane 35 pills are classified as oral contraceptives, which effectively reduces circulating androgens and are treatment for hyperandrogenism caused androgenic skin symptoms and irregular menstrual cycles. GLP-1 Receptor Agonist(e.g. exenatide, liraglutide) have the effects of lowering blood sugar and weight control by inhibiting of gastric emptying and reducing food intake. This study aims to evaluate the effect of metformin-GLP-1 Receptor agonist combination versus metformin-Diane-35 combination treatment on lipid metabolism and cardiovascular risks in overweight polycystic ovarian syndrome (PCOS) patients.

DETAILED DESCRIPTION:
Groups:

Experimental treatment: Metformin-GLP-1 Receptor Agonist Therapy.

Regular treatment: Metformin-Oral Contraceptive(OC) Therapy.

Time Point:

Initial treatment;

Post-treatment (4w);

Post-treatment (8w);

Post-treatment (12w);

Assess reproductive functions and cardiovascular risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of PCOS according to the Rotterdam criteria based on the presence of two of three criteria: oligomenorrhoea, clinical or biochemical hyperandrogenism and polycystic ovaries on ultrasound after exclusion of other endocrine causes of hyperandrogenism.
* Participants had no concurrent illness and were not on any prescription or over-the-counter medication that was likely to affect insulin sensitivity or lipids for the preceding 12 weeks.
* Participants were advised not to change physical activity or dietary habits during the study period. All subjects were overweight/obese [body mass index (BMI) >=24 kg/m2 or waistline>=85cm ].
* All subjects had normal thyroid-stimulating hormone and prolactin levels.

Exclusion Criteria:

* smoking, alcohol use, or having taken medication within 2 months of the study that is known to affect reproductive or metabolic functions.
* age below 18 yr or over 50 yr.
* postmenopausal.
* uncontrolled hypertension (blood pressure >=160/100 mm Hg).
* preexisting OPs or GLP-1 agonists supplementation
* alcohol intake greater than 20 g/d, or pregnancy.
* signs of liver or renal failure or active liver disease (ALT > 2.5× the upper limit of normal values).
* PLT<60*10^9/L,Hb<100g/L, smoking, alcohol use.
* The patient that cannot complete the intervention or have other conditions that is not appropriate to enter the group, such as patients who are taking glucocorticoid steroids or malignant tumor treatment, etc.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Min long, MD, Principal Investigator — Department of Endocrinology, Xinqiao Hospital,Third Military Medical University
Locations (1):
- The Second Affiliated Hospital, Third Military Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be avaliable within 6 months of study completion.
Access Criteria: Data access requests will be reviewed by an external independent review panel. Requestors will be required to sign a data access agreement.
URL: http://bethesda.org

REFERENCES:
- [Result] Macut D, Bjekic-Macut J, Rahelic D, Doknic M. Insulin and the polycystic ovary syndrome. Diabetes Res Clin Pract. 2017 Aug;130:163-170. doi: 10.1016/j.diabres.2017.06.011. Epub 2017 Jun 12. PMID 28646699
- [Result] Zhou BF; Cooperative Meta-Analysis Group of the Working Group on Obesity in China. Predictive values of body mass index and waist circumference for risk factors of certain related diseases in Chinese adults--study on optimal cut-off points of body mass index and waist circumference in Chinese adults. Biomed Environ Sci. 2002 Mar;15(1):83-96. PMID 12046553
- [Result] Barthelmess EK, Naz RK. Polycystic ovary syndrome: current status and future perspective. Front Biosci (Elite Ed). 2014 Jan 1;6(1):104-19. doi: 10.2741/e695. PMID 24389146
- [Result] Dumesic DA, Oberfield SE, Stener-Victorin E, Marshall JC, Laven JS, Legro RS. Scientific Statement on the Diagnostic Criteria, Epidemiology, Pathophysiology, and Molecular Genetics of Polycystic Ovary Syndrome. Endocr Rev. 2015 Oct;36(5):487-525. doi: 10.1210/er.2015-1018. PMID 26426951
- [Result] Rotterdam ESHRE/ASRM-Sponsored PCOS consensus workshop group. Revised 2003 consensus on diagnostic criteria and long-term health risks related to polycystic ovary syndrome (PCOS). Hum Reprod. 2004 Jan;19(1):41-7. doi: 10.1093/humrep/deh098. PMID 14688154
- [Result] Yildiz BO, Bozdag G, Yapici Z, Esinler I, Yarali H. Prevalence, phenotype and cardiometabolic risk of polycystic ovary syndrome under different diagnostic criteria. Hum Reprod. 2012 Oct;27(10):3067-73. doi: 10.1093/humrep/des232. Epub 2012 Jul 9. PMID 22777527
- [Result] Farrell K, Antoni MH. Insulin resistance, obesity, inflammation, and depression in polycystic ovary syndrome: biobehavioral mechanisms and interventions. Fertil Steril. 2010 Oct;94(5):1565-74. doi: 10.1016/j.fertnstert.2010.03.081. Epub 2010 May 14. PMID 20471009
- [Result] Escobar-Morreale HF. Polycystic ovary syndrome: definition, aetiology, diagnosis and treatment. Nat Rev Endocrinol. 2018 May;14(5):270-284. doi: 10.1038/nrendo.2018.24. Epub 2018 Mar 23. PMID 29569621
- [Result] Ruan X, Kubba A, Aguilar A, Mueck AO. Use of cyproterone acetate/ethinylestradiol in polycystic ovary syndrome: rationale and practical aspects. Eur J Contracept Reprod Health Care. 2017 Jun;22(3):183-190. doi: 10.1080/13625187.2017.1317735. Epub 2017 May 2. PMID 28463030
- [Result] Wang YW, He SJ, Feng X, Cheng J, Luo YT, Tian L, Huang Q. Metformin: a review of its potential indications. Drug Des Devel Ther. 2017 Aug 22;11:2421-2429. doi: 10.2147/DDDT.S141675. eCollection 2017. PMID 28860713
- [Result] Jiang Y, Wang Z, Ma B, Fan L, Yi N, Lu B, Wang Q, Liu R. GLP-1 Improves Adipocyte Insulin Sensitivity Following Induction of Endoplasmic Reticulum Stress. Front Pharmacol. 2018 Oct 16;9:1168. doi: 10.3389/fphar.2018.01168. eCollection 2018. PMID 30459598
- [Derived] Liao M, Li X, Zhang H, Zhou L, Shi L, Li W, Shen R, Peng G, Zhao H, Shao J, Wang X, Sun Z, Zheng H, Long M. Effects and plasma proteomic analysis of GLP-1RA versus CPA/EE, in combination with metformin, on overweight PCOS women: a randomized controlled trial. Endocrine. 2024 Jan;83(1):227-241. doi: 10.1007/s12020-023-03487-4. Epub 2023 Aug 31. PMID 37653215

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Metformin-GLP-1 Receptor Agonist | Metformin-Oral Contraceptive(OC)
Started | 35 | 35
Completed | 30 | 30
Not Completed | 5 | 5
Not completed — Lost to Follow-up | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metformin-Oral Contraceptive(OC) | Metformin-GLP-1 Receptor Agonist | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7 | 3 | 10
  Between 18 and 65 years | 23 | 27 | 50
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.43 (5.30) | 25.73 (4.95) | 24.08 (5.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 30 | 60
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  China | 30 | 30 | 60
weight [Mean (Standard Deviation); unit: kg] | 70.98 (11.02) | 73.95 (10.04) | 72.47 (10.56)

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Reproductive Functions
Description: Concentration of LH was measured in mIU/ml.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: mIU/ml
Arm/Group | Metformin-GLP-1 Receptor Agonist | Metformin-Oral Contraceptive(OC)
Number analyzed (Participants) | 30 | 30
mIU/ml | 5.52 (3.37) | 5.33 (2.52)

2. Secondary Outcome: Basic Vital Signs
Description: Weight and height will be combined to report BMI in kg/m^2.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Metformin-GLP-1 Receptor Agonist | Metformin-Oral Contraceptive(OC)
Number analyzed (Participants) | 30 | 30
kg/m^2 | 26.26 (3.67) | 27.12 (4.04)

3. Secondary Outcome: Assessment of Liver Function
Description: Alanine transaminase was measured in IU/L.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Metformin-GLP-1 Receptor Agonist | Metformin-Oral Contraceptive(OC)
Number analyzed (Participants) | 30 | 30
IU/L | 39.09 (24.16) | 36.73 (43.12)

4. Secondary Outcome: Assessment of Blood Pressure
Description: Systolic blood pressure was measured in mmHg.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Metformin-GLP-1 Receptor Agonist | Metformin-Oral Contraceptive(OC)
Number analyzed (Participants) | 30 | 30
mmHg | 122.83 (10.91) | 122.40 (6.39)

5. Secondary Outcome: Assessment of Reproductive Function
Description: Changes in testosterone levels were measured
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Metformin-GLP-1 Receptor Agonist | Metformin-Oral Contraceptive(OC)
Number analyzed (Participants) | 30 | 30
nmol/L | 1.82 (0.51) | 2.14 (1.02)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Metformin-GLP-1 Receptor Agonist | Metformin-Oral Contraceptive(OC)
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 1/30
OTHER ADVERSE EVENTS (reported when occurring in more than 3.33% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin-GLP-1 Receptor Agonist (N=30) | Metformin-Oral Contraceptive(OC) (N=30)
Aminopherase elevation (Hepatobiliary disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Limitations of this trial include a relatively small sample size and single-center design.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-07-28): https://cdn.clinicaltrials.gov/large-docs/05/NCT03151005/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-28): https://cdn.clinicaltrials.gov/large-docs/05/NCT03151005/SAP_001.pdf